# **INFORMED CONSENT FORM (ICF)**

**Official Title:** The Impact of Stationary Combined Exercise on Adiponectin and High-Sensitivity C-Reactive Protein Levels in Overweight Women

NCT Number: NCT number pending

**Document Type:** Informed Consent Form (Final Version)

Document Date: January 15, 2024

Version: v1.0

**Institution:** College of Physical Education and Health, Chongqing College of International Business and Economics, Hechuan, Chongqing, China

#### 1. Introduction

You are invited to participate in a research study conducted by Prof. Xianjie Zheng at the College of Physical Education and Health, Chongqing College of International Business and Economics. Before deciding to participate, please read this form carefully. It explains the purpose of the study, what will happen if you participate, possible risks and benefits, and your rights as a volunteer.

### 2. Purpose of the Study

The purpose of this research is to study the effects of an eight-week program of stationary combined (circuit) exercise on levels of adiponectin and high-sensitivity C-reactive protein (hs-CRP) in overweight young women. These biomarkers are related to inflammation and cardiovascular health. The study aims to understand how exercise can improve these factors.

#### 3. Procedures

If you agree to participate, you will be randomly assigned to either an exercise group or a control group. The exercise group will participate in four exercise sessions each week for eight weeks. Each session will include warm-up, circuit-based exercises (such as sit-ups, push-ups, step jumps, and jump rope), and cool-down. Exercise intensity will be maintained at 70–90% of your maximum heart rate and will be supervised by trained researchers. Blood samples will be collected before and 48 hours after the last exercise session to measure levels of adiponectin and hs-CRP using ELISA kits. Your body composition (weight, body fat percentage, and BMI) and VOmmax will also be measured.

#### 4. Duration

Participation in this study will last approximately 8 weeks, including initial screening, training, and follow-up testing.

### 5. Risks and Discomforts

The study involves minimal risks. You may experience temporary muscle soreness, fatigue, or shortness of breath during exercise sessions. All exercise sessions will be supervised by qualified personnel, and safety measures will be in place. Blood sampling may cause minor discomfort or bruising at the puncture site. If you feel unwell during the sessions, you should immediately inform the researcher and stop the activity.

### 6. Potential Benefits

While you may not directly benefit from participating, your involvement may improve your physical fitness, cardiovascular health, and overall well-being. The study's results may help researchers and health professionals design better exercise programs to improve metabolic health in overweight women.

## 7. Confidentiality

All personal information collected during this study will remain strictly confidential. Your name will not appear in any reports or publications. Data will be coded and stored securely, accessible only to the research team. ClinicalTrials.gov and the institutional ethics committee may review the anonymized data for verification.

### 8. Voluntary Participation and Withdrawal

Your participation in this study is entirely voluntary. You may refuse to participate or withdraw at any time without any penalty or loss of benefits. Your decision will not affect your relationship with the university or any of its programs. If you decide to withdraw, all collected data will be destroyed upon your request unless already anonymized.

### 9. Compensation

You will not receive financial compensation for participating in this study. However, the study will cover any costs associated with laboratory testing or exercise supervision.

### 10. Contacts

If you have any questions about this research, please contact: **Principal Investigator:** Prof. Xianjie Zheng College of Physical Education and Health, Chongqing College of International Business and Economics, Hechuan, Chongqing, China Email: xianjiezheng1@gmail.com Phone: +86-23-62893102 If you have questions about your rights as a research participant, you may contact the institutional ethics committee at the same address.

### 11. Consent Statement

By signing below, you acknowledge that you have read and understood the information provided above. You have had the opportunity to ask questions and have received satisfactory answers. You voluntarily agree to participate in this study.

| Participant's | Name: | Date: | Signature: |
|----------------|-------|-----------|------------|
| Investigator's | Name: | <br>Date: | Signature: |

#### End of Document